CLINICAL TRIAL: NCT05156008
Title: Comparison of Ultrasound-guided and Palpation-inserted Peripheral Venous Cannula in Patients Before Primary Hip or Knee Arthroplasty a Randomized Controlled Trial
Brief Title: Comparison of Ultrasound-guided and Palpation-inserted Peripheral Venous Cannula
Acronym: CompOne
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica (Other)
Responsible Party: Principal Investigator, Jakub Hlasny, MD, EDRA, Principal investigator, F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 26/2021
Record Dates: First submitted 2021-09-15; First posted 2021-12-14 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Vascular Access Complication; Vascular Access Site Bruising
Keywords: Ultrasound-guided vascular access; Randomized trial; Vascular access

STUDY DESIGN:
Intervention Model Description: Comparison of two arms. One arm ultrasound guided vascular access (UGVA) and control group standard vein cannulation with palpation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (No Intervention): Patient on the operating room, before primary hip or knee arthroplasty, will have his or her cannula inserted by standard palpation of vein under strict aseptic measures. Application of tourniquet on upper arm, palpation of vein, disinfection of skin and insertion of cannula. After two unsuccessful punctures, UGVA operator will step in and perform insertion of cannula with ultrasound.
  Medical staff will note:
  * number of attempts
  * time to obtain vascular access
  * type of cannula
  * DIVA score
- Group B (Other): Patient on the operating room, before primary hip or knee arthroplasty, will have his or her cannula inserted by ultrasound guided vascular access under strict aseptic measures. With or without tourniquet applied on upper arm operator will prescan vasculature of arm to choose applicable vein. After disinfection of skin optimal vein is on plain part of arm and cannula must not end in flection (elbow, wrist) of arm.
  Medical staff will note:
  * number of attempts, if 2 attempts fail, another operator will perform insertion
  * time to obtain vascular access
  * diameter of vein
  * type of cannula
  * DIVA score
  Interventions: Other: Ultrasound-guided vascular access

INTERVENTIONS:
Other: Ultrasound-guided vascular access — Patients in this arm will have peripheral venous cannula inserted under realtime ultrasound guidance. Out of plane technique (in plane technique if too deep when tip of the needle is on vessel wall) used by experienced physicians in UGVA. Out of plane technique strictly used in step by step manner. That means moving probe with the tip of the needle to always locate its exact position, all the way into the vein. All performed insertions are carried out by skilled operators in UGVA with out of plane technique. Just before surgery in block room.
  Arms: Group B

SUMMARY:
Every patient need venous access for surgery under anesthesia. It is the most frequently performed invasive procedure in medicine in the whole world. In expert groups, ultrasonographically guided vascular access (UGVA) appears to be a significantly better method, but studies on larger groups of patients are lacking.

Prospective randomized 2-arm study which is comparing success rate of ultrasound guided a palpation inserted cannulas in patients undergoing primary hip or knee arthroplasty.

The project will be managed according to the protocol of principles of Good Clinical Practice and valid regulations.

DETAILED DESCRIPTION:
More than 2 billion peripheral vascular cannulas (PVCs) are introduced globally each year. Each patient needs venous access for surgery under anesthesia. It is the most frequently performed invasive procedure in medicine in the whole world. Nevertheless, investigators still do not know how to fix them adequately, to work reliably for at least 72 hours.

Then there is a group of patients with difficult intravenous access (DIVA). These patients often have to undergo repeated painful punctures through the skin when introducing PVC. Many times well trained healthcare worker in the ultrasound-guided vascular access is needed to introduce PVC in DIVA patients. Up to one third of adult patients are DIVA. In overweight orthopedic patients, this subpopulation can reach up to 50% . Up to 64% PVC fails within 72 hours.

Several studies have shown that PVC introduced at the site of limb flexion (elbow, wrist), repeated punctures increase the risk of thrombosis, infection and phlebitis. In expert groups, ultrasonographically guided vascular access (UGVA) appears to be a significantly better method, but studies on larger groups of patients are lacking.

Investigators hypothesise that UGVA is superior in many parameters. The aim of our study is to compare two types of cannula insertion methods and their benefits and risks for patients. Ultrasound guided insertion and palpation guided insertion. To have evidence robust enough and after statistical analysis investigators decided for sample of 500 patients.

Investigators will evaluate data after 100, 250 and 500 patients. After statistical analysis will be calculate benefit/risk ratio for patients and take steps towards patient safety and satisfaction.

The project will be managed according to the protocol of principles of Good Clinical Practice and valid regulations.

Patients are divided in two groups. Group A (insertion by palpation of vein): standard cannula (name brand "vasofix" BBraun) insertion through vein palpation and insertion in block room.

- prior insertion medical staff will fill in study protocol form A

Group B (UGVA): DIVA score calculation, Ultrasound-guided (name brand "deep access introcan" BBraun) cannula insertion

- prior insertion medical staff will fill in study protocol form B

In primary outcome investigators hypothesised that UGVA need less attempts to successful cannulation in comparison with vein cannulation by palpation. Investigators also think that deep vein cannula secured by UGVA will have lower failure rates by any means. In general there are several benefits in UGVA. On the other hand all above is applicable only in hands of well trained medical staff.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip or knee arthroplasty
* BMI over 25

Exclusion Criteria:

* reoperation of endoprosthesis
* mental disorder
* age under 18
* sepsis
* protocol non-compliance
* gravidity
* patient refusal or no informed consent or both

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Ultrasound guided venous access need less attempts to successful cannulation | up to 24 hours
  Number of punctures through skin defines number of attempts. Every puncture of skin with cannula is considered as attempt. Number of attempts are recorded in protocol as whole number. Does not matter with technique is used.

SECONDARY OUTCOMES:
Ultrasound guided venous access time to successful cannulation | up to 24 hours
  Time measurement starts when operator puts probe on patient and starts prescan of veins. Time measurement stops when cannula is successfully inserted confirmed by blood return after removal of internal metal piece. Is measured in minutes and seconds.
Venous access by palpation time to successful cannulation | up to 24 hours
  Time measurement starts when nurse or physician starts to assess veins. Tourniquet application, disinfection of skin, palpation and cannulation are considered as process of cannulation. Time measurement stops when cannula is successfully inserted confirmed by blood return after removal of internal metal piece. Is measured in minutes and seconds.
Ultrasound guided venous access allows insertion of cannulas suitable for blood drawing | up to 5 days
  During UGVA measurement of vein diameter measurement is mandatory. If diameter of vein in millimeters is equal to higher to Fr of catheter/cannula it should allow to draw blood without need for repeated vein punctures for blood sampling. Cannula G22 need 2,7mm vein diameter, Cannula G20 need 3,3mm vein diameter. Cannula G18 need 3,9mm vein diameter. In protocol there is mark on every day that cannula allows blood drawing. Is marked as yes-no immediately after insertion, and than every day until removal of cannula.
UGVA will reduce the costs associated with perioperative venous access | up to 5 days
  In protocol there is mark for every material associated with blood drawing, venous access. After 5 days there will be sum of cost of material used. Up to 5 days or patient discharge.
Cannulas suitable for blood drawing, shortens the time a nurse spends drawing blood in the postoperative period at the ward | up to 5 days
  Every need of blood draw is marked in protocol, time spend to draw blood is marked in protocol. Measured in minutes and seconds. There are to scenarios. Blood draw through cannula: Measurement starts the moment nurse applies flush of saline, after that nurse will draw blood according to protocol, time measurement stops when saline flush is administered after successful blood draw. If not successful then measurement continues through blood draw by venipuncture.
  Scenario two: blood draw through venipuncture: time measurement starts when nurse starts to assess veins for venipuncture. Time measurement stops after successful blood draw and after venipuncture site covering with tampon and tape.
Insertion site infection occurrence after cannula placement | up to 5 days
  In protocol there is mark using "madonn scale - peripheral cannulas site infection 0 - 4" for every day in cannula is in use
Long peripheral venous cannulas inserted under ultrasound guidance have low failure rate for intravenous therapy | through study completion, an average of 1 year
  Inability to administer intravenous therapy through cannula from any reason is considered as failure of cannula. Failure rate is calculated from ratio of cannulas that did not fail to cannulas that failed. Is marked in results as percentage (%) as whole number and two decimals.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Hlasny, MD, Principal Investigator — physician of anesthesia and intensive care department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Witting MD. IV access difficulty: incidence and delays in an urban emergency department. J Emerg Med. 2012 Apr;42(4):483-7. doi: 10.1016/j.jemermed.2011.07.030. Epub 2011 Dec 2. PMID 22137793
- [Result] Alexandrou E, Ray-Barruel G, Carr PJ, Frost S, Inwood S, Higgins N, Lin F, Alberto L, Mermel L, Rickard CM. International prevalence of the use of peripheral intravenous catheters. J Hosp Med. 2015 Aug;10(8):530-3. doi: 10.1002/jhm.2389. Epub 2015 Jun 3. PMID 26041384
- [Result] Ahlqvist M, Berglund B, Nordstrom G, Klang B, Wiren M, Johansson E. A new reliable tool (PVC assess) for assessment of peripheral venous catheters. J Eval Clin Pract. 2010 Dec;16(6):1108-15. doi: 10.1111/j.1365-2753.2009.01278.x. PMID 19925593
- [Result] Webster J, Clarke S, Paterson D, Hutton A, van Dyk S, Gale C, Hopkins T. Routine care of peripheral intravenous catheters versus clinically indicated replacement: randomised controlled trial. BMJ. 2008 Jul 8;337(7662):a339. doi: 10.1136/bmj.a339. PMID 18614482
- [Derived] Hlasny J, Alberty R, Hlavac M, Grgac I, Grey MT, Venglarcik M. Comparison of ultrasound-guided and palpation-inserted peripheral venous cannula in -patients before primary hip or knee arthroplasty: study protocol for a randomized controlled trial. Trials. 2023 Jul 21;24(1):467. doi: 10.1186/s13063-023-07459-x. PMID 37480132